CLINICAL TRIAL: NCT02721524
Title: Comparison Between Outcomes Of Ring And Suture Annuloplasty For Functional Tricuspid Regurgitation In Rheumatic Mitral Valve Diseases
Brief Title: Ring Versus Suture Annuloplasty For Functional Tricuspid Regurgitation In Rheumatic Mitral Valve Diseases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Gangalal National Heart Centre (Other)
Responsible Party: Principal Investigator, Marisha Aryal, Resident, Cardiac Surgery Dept., Shahid Gangalal National Heart Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRICUSPID STUDY-RCT
Record Dates: First submitted 2016-03-16; First posted 2016-03-29 (Estimated); Last update posted 2016-03-29 (Estimated); Status verified 2016-03

CONDITIONS: Functional Tricuspid Regurgitation
Keywords: Ring Annuloplasty; Suture Annuloplasty; Functional Tricuspid Regurgitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group R (ring) (Active Comparator): Patients in Group R will undergo tricuspid ring annuloplasty
  Interventions: Procedure: Tricuspid Annuloplasty
- Group S (suture) (Active Comparator): Patients in Group S will undergo De Vega's suture annuloplasty
  Interventions: Procedure: Tricuspid Annuloplasty

INTERVENTIONS:
Procedure: Tricuspid Annuloplasty — Patients will undergo repair of tricuspid regurgitation

SUMMARY:
This study aims to compare whether De Vega's Suture annuloplasty is equally effective in reducing the progression of Functional Tricuspid regurgitation as that claimed for Ring annuloplasty in Rheumatic Heart Disease patients with concurrent Mitral valve replacement.

DETAILED DESCRIPTION:
Functional Tricuspid regurgitation (FTR) occurs due to annular dilatation in association with left sided valve disease and is more commonly seen than primary pathology in patients with Rheumatic mitral valve disease. FTR occurs due to increased right ventricle after load that leads to either dilatation or geometric deformation of Tricuspid annulus. If left untreated, FTR may worsen and increase morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* The participants will be all patients between 15 to 75 years of age group diagnosed as a case of Rheumatic Mitral Valve disease with moderate to severe functional Tricuspid regurgitation.

Exclusion Criteria:

* Patient with organic Tricuspid Valve (TV) lesion diagnosed in Echocardiography
* Patient with FTR requiring Mitral Valve repair
* Patient with FTR requiring concomitant aortic valve replacement
* Patient with FTR secondary to pathology other than Mitral valve disease

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Improvement in severity of FTR | within 3 months
  Definitions:
  1. Improvement in FTR: refers to Mild or No TR
  2. Tricuspid regurgitation is graded as mild, moderate, and severe based on regurgitant jet area i. <5cm2 = Mild ii. 6-10cm2 = Moderate iii. >10cm2 = Severe

SECONDARY OUTCOMES:
Mortality | up to 3 months of intervention
  Mortality: Mortality within hospital stay or 3 months postoperative.

CONTACTS AND LOCATIONS:
Overall Officials: Marisha Aryal, MBBS, Principal Investigator — Shahid Gangalal National Heart Centre
Locations (1):
- Shahid Gangalal National Heart Centre, Kathmandu, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tang GH, David TE, Singh SK, Maganti MD, Armstrong S, Borger MA. Tricuspid valve repair with an annuloplasty ring results in improved long-term outcomes. Circulation. 2006 Jul 4;114(1 Suppl):I577-81. doi: 10.1161/CIRCULATIONAHA.105.001263. PMID 16820641
- [Background] Guenther T, Mazzitelli D, Noebauer C, Hettich I, Tassani-Prell P, Voss B, Lange R. Tricuspid valve repair: is ring annuloplasty superior? Eur J Cardiothorac Surg. 2013 Jan;43(1):58-65; discussion 65. doi: 10.1093/ejcts/ezs266. Epub 2012 May 24. PMID 22627660
- [Background] Sarralde JA, Bernal JM, Llorca J, Ponton A, Diez-Solorzano L, Gimenez-Rico JR, Revuelta JM. Repair of rheumatic tricuspid valve disease: predictors of very long-term mortality and reoperation. Ann Thorac Surg. 2010 Aug;90(2):503-8. doi: 10.1016/j.athoracsur.2010.03.105. PMID 20667339
- [Background] Rivera R, Duran E, Ajuria M. Carpentier's flexible ring versus De Vega's annuloplasty. A prospective randomized study. J Thorac Cardiovasc Surg. 1985 Feb;89(2):196-203. PMID 3881631
- [Background] Badano LP, Muraru D, Enriquez-Sarano M. Assessment of functional tricuspid regurgitation. Eur Heart J. 2013 Jul;34(25):1875-85. doi: 10.1093/eurheartj/ehs474. Epub 2013 Jan 9. PMID 23303656
- [Result] Rogers JH, Bolling SF. The tricuspid valve: current perspective and evolving management of tricuspid regurgitation. Circulation. 2009 May 26;119(20):2718-25. doi: 10.1161/CIRCULATIONAHA.108.842773. PMID 19470900
- [Result] McCarthy PM, Bhudia SK, Rajeswaran J, Hoercher KJ, Lytle BW, Cosgrove DM, Blackstone EH. Tricuspid valve repair: durability and risk factors for failure. J Thorac Cardiovasc Surg. 2004 Mar;127(3):674-85. doi: 10.1016/j.jtcvs.2003.11.019. PMID 15001895
- [Result] Navia JL, Nowicki ER, Blackstone EH, Brozzi NA, Nento DE, Atik FA, Rajeswaran J, Gillinov AM, Svensson LG, Lytle BW. Surgical management of secondary tricuspid valve regurgitation: annulus, commissure, or leaflet procedure? J Thorac Cardiovasc Surg. 2010 Jun;139(6):1473-1482.e5. doi: 10.1016/j.jtcvs.2010.02.046. Epub 2010 Apr 14. PMID 20394950